CLINICAL TRIAL: NCT00044824
Title: A Multicenter, Double-Blind, Randomized, Parallel Groups Placebo-Controlled Study to Assess the Efficacy and Safety of Fexofenadine 120mg BID in Subjects With Mild to Moderate Persistent Asthma
Brief Title: Efficacy and Safety of Fexofenadine in Mild to Moderate Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M016455P/3002; M016455
Record Dates: First submitted 2002-09-05; First posted 2002-09-17 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fexofenadine

INTERVENTIONS:
Drug: Fexofenadine

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of fexofenadine 120mg BID compared to placebo in the treatment of subjects with mild to moderate persistent asthma

DETAILED DESCRIPTION:
The incidence of respiratory allergy in the US has increased gradually over the past several years, and current estimates suggest that allergic rhinitis and bronchial asthma affect approximately 20% and 5% of the population, respectively. Rhinitis and asthma frequently coexist, and large-scale population surveys indicate that up to 38% of subjects with rhinitis have asthma, and up to 78% of subjects with asthma have chronic nasal symptoms. Safety concerns with the increased use of inhaled corticosteroids, the heterogeneity of the disease, and poor compliance with asthma medication regimens, point to the need for the development of safe and convenient oral therapies for asthma. Histamine is an important chemical mediator of inflammation in asthma. The benefits of antihistamine treatment in patients with mild to moderate asthma have been well documented, however their clinical use has been previously limited due to the high doses required for efficacy and their associated side effects including sedation and cognitive impairment.

Recent evidence indicates that in addition to H1-receptor antagonism, some of the newer nonsedating, non-impairing antihistamines appear to possess various anti-inflammatory properties at concentrations achieved at therapeutic dosages suggesting an additional benefit of these drugs in the management of allergic diseases and asthma. The purpose of this study is to investigate the efficacy and safety of fexofenadine 120mg BID compared to placebo in the treatment of subjects with mild to moderate persistent asthma.

ELIGIBILITY:
Inclusion criteria:

* Males and non-pregnant, non-breastfeeding females 12 through 80 years of age
* FEV1 in the context of this study is greater than 60% and not less or equal to 87% of predicted values at Visit 1 or Visit 2 (and no short-acting agent beta-agonist use within 6 hours prior to spirometry)
* Improvement in FEV1 of at least 12% of predicted value and at least 200ml within 15 to 30 minutes of inhaling 2 puffs of albuterol 90mcg/actuation demonstrated at study entry OR documented during the previous 12 months at the study site.
* Use of a short-acting, beta-agonist inhaler to treat asthma symptoms on an average of at least 2 days per week during the previous 2 weeks (greater than or equal to 4 days total during the previous 2 weeks, excluding prophylactic use).

Exclusion criteria:

* Otherwise healthy

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2002-02; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Forced Expiratory Volume FEV1

SECONDARY OUTCOMES:
Change in Daily Asthma Symptoms Score from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (7):
- Aventis Pharmaceuticals Inc., Bridgewater, New Jersey, United States
- Sanofi-Aventis Admnistrative Office, Costa Rica, Costa Rica
- Sanofi-Aventis Administrative Office, Guatemala City, Guatemala
- sanofi-aventis Hungaria, Budapest, Hungary
- Sanofi-Aventis Administrative Office, México, Mexico
- sanofi-aventis Poland, Warsaw, Poland
- Sanofi-Aventis Aministrative Office, Moscow, Russia

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com